CLINICAL TRIAL: NCT02005484
Title: An Open-label Pilot Study of Herceptin Monotherapy on Objective Treatment Response in Patients With Metastatic or Locally Advanced Gastric Cancer Who Had Disease Progression During Platinum-based or 5-fluoropyrimidine-based Chemotherapy
Brief Title: A Study of Herceptin (Trastuzumab) in Patients With Metastatic or Advanced Gastric Cancer With Disease Progression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to slow patient recruitment.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17263
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab

ARMS (1):
- Trastuzumab Monotherapy (Experimental): Initial dose of 4 milligrams (mg) per (/) kilogram (kg) by body weight (BW), followed by 2 mg/kg BW at each subsequent visit
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — 4 mg/kg initial dose, followed by 2 mg/kg
  Other Names: Herceptin

SUMMARY:
This study will evaluate the efficacy and safety of Herceptin in patients with metastatic or advanced gastric cancer with disease progression during platinum-based or 5-fluoropyrimidine-based chemotherapy. The anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-75 years of age;
* metastatic or advanced gastric cancer;
* disease progression under or after 1 prior platinum-based or 5-fluoropyrimidine-based chemotherapy for metastatic disease;
* >=4 weeks from last platinum-based or fluoropyrimidine-based chemotherapy;
* >=1 measurable lesion;
* HER2 overexpression (IHC [2+] or [3+]).

Exclusion Criteria:

* concurrent chemotherapy or immunotherapy;
* brain or meningeal metastases;
* clinically significant cardiac disease, advanced pulmonary disease or severe dyspnoea;
* co-existing malignancies or malignancies diagnosed within last 5 years, except basal cell cancer or cervical cancer in situ;
* women who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (11):
- Vienna, Austria
- Germany (10):
  - Dresden
  - Erlangen
  - Essen
  - Grenzach-Wyhlen
  - Halle
  - Kassel
  - Kiel
  - Mannheim
  - München
  - Oldenburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab Monotherapy: Participants received trastuzumab at an initial dose of 4 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1, followed by maintenance doses of 2 mg/kg, IV, once weekly starting on Day 8 up to a maximum of 33 weeks.
Period: Overall Study
Arm/Group | Trastuzumab Monotherapy
Started | 6
Completed | 2
Not Completed | 4
Not completed — Death | 1
Not completed — Disease progression | 1
Not completed — Changed to a Different Study | 1
Not completed — Sponsor decision | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all participants who signed informed consent for the study.
Groups:
- Trastuzumab Monotherapy: Participants received trastuzumab at an initial dose of 4 mg/kg IV on Day 1, followed by maintenance doses of 2 mg/kg, IV, once weekly starting on Day 8 up to a maximum of 33 weeks.
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.49 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response by Response Evaluation Criteria In Solid Tumors (RECIST) Category
Description: Tumor response assessed according to RECIST. Complete response (CR): complete disappearance of all target and non-target lesions, with exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<]10 millimeters [mm]); no new lesions. Partial response (PR): greater than or equal to (≥)30 percent (%) decrease under baseline of sum of diameters of all target lesions. Short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions; no unequivocal progression of non-target disease; no new lesions. Stable disease (SD): not qualifying for CR, PR, or progressive disease (PD). Participants who could not be classified per RECIST were allocated as follows: early death from malignant disease (death due to cancer), early death because of other cause (death not related to toxicity or cancer disease), and unknown (for not fitting into the above categories).
Time Frame: Weekly throughout study
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
percentage of participants
  CR | 0
  PR | 33.3
  SD | 0
  PD | 50.0
  Early death from malignant disease | 0
  Early death because of other cause | 16.7
  Unknown | 0

2. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Participants were classified as having a clinical benefit if they had a best overall tumor response of CR, PR, or SD. Tumor response assessed according to RECIST. CR: complete disappearance of all target and non-target lesions, with exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm); no new lesions. PR: ≥30% decrease under baseline of sum of diameters of all target lesions. Short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions; no unequivocal progression of non-target disease; no new lesions. Stable SD: not qualifying for CR, PR, or PD.
Time Frame: Weekly throughout the study
Population: ITT population
Measure: Number; unit: percentage participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
percentage participants | 33.3

3. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR or PR
Description: Tumor response assessed according to RECIST. CR: complete disappearance of all target and non-target lesions, with exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm); no new lesions. PR: ≥30% decrease under baseline of sum of diameters of all target lesions. Short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions; no unequivocal progression of non-target disease; no new lesions.
Time Frame: Weekly throughout the study
Population: ITT population
Measure: Number; unit: percentage participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
percentage participants | 33.3

4. Secondary Outcome: Overall Survival - Number of Participants Who Died
Description: OS was defined as the time, in months, from the date of study entry to the date of the death due to any cause. If a participant's date of death was unknown, or had not occurred, the last date of examination, treatment, and follow-up dates were included in the analysis.
Time Frame: Weekly throughout the study
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
participants | 2

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time, in months, from the date of study entry to the date of the death due to any cause. If a participant's date of death was unknown, or had not occurred, the last date of examination, treatment, and follow-up dates were included in the analysis.
Time Frame: Weekly throughout the study
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
months | 6.39 [1.4 to 18.7]

6. Secondary Outcome: Time to Progression - Number of Participants With an Event
Description: Time to progression was defined as the time, in months, from the date of study entry to the date of disease progression or death due to any cause. If a participant's date of disease progression or death was unknown, or had not occurred, the last date of examination, treatment, and follow-up dates were included in the analysis.
Time Frame: Weekly throughout the study
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
participants | 5

7. Secondary Outcome: Time to Progression
Description: as for outcome 6
Time Frame: Weekly throughout the study
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Trastuzumab Monotherapy
Number analyzed (Participants) | 6
months | 1.78 [1.4 to 7.4]

ADVERSE EVENTS:
Time Frame: Weekly throughout the study.
Description: All participants who received at least 1 dose of study treatment were included in the safety analysis population.
Groups:
- Trastuzumab Monotherapy: Participants received trastuzumab via IV infusion once weekly at an initial dose of 4 mg/kg at Visit 1, and 2 mg/kg at each subsequent visit for a maximum of 33 visits.
Arm/Group | Trastuzumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Monotherapy (N=6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Stent placement (Surgical and medical procedures) | 1
Oesophageal stent insertion (Surgical and medical procedures) | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1
Hypersensitivity (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Monotherapy (N=6)
Abdominal pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Retching (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Oesophageal fistula (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 1
Hyperhidrosis (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Onychomycosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Stent removal (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to slow patient recruitment, the study was prematurely terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.